CLINICAL TRIAL: NCT05949242
Title: Comparison of Clinical Outcomes in Patients Undergoing Cataract Surgery With OMNI Canaloplasty vs Cataract Surgery With OMNI Canaloplasty and Hydrus Stent
Brief Title: Clinical Outcomes in Cataract Surgery With OMNI Canaloplasty vs Cataract Surgery With OMNI Canaloplasty and Hydrus Stent
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ridge Eye Care (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Douglas McGraw, D.O., Principal Investigator, Ridge Eye Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 76998263
Record Dates: First submitted 2023-07-10; First posted 2023-07-17 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Participants will have one eye randomized to each arm of the trial:
  one eye will receive OMNI canaloplasty alone the other eye will receive OMNI canaloplasty and Hydrus microstent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- OMNI canaloplasty with cataract surgery (Active Comparator): participant will undergo OMNI canaloplasty with cataract surgery in one randomized eye
  Interventions: Device: OMNI canaloplasty
- OMNI canaloplasty and Hydrus with cataract surgery (Active Comparator): participant will undergo OMNI canaloplasty and Hydrus with cataract surgery in the contralateral eye
  Interventions: Device: OMNI canaloplasty; Device: Hydrus microstent

INTERVENTIONS:
Device: OMNI canaloplasty — OMNI device is used to catheterize Schlemm's canal for 180 degrees and perform canaloplasty. Viscoelastic is eluded upon retraction of the catheter performing viscodilation of the canal
Device: Hydrus microstent — Hydrus stent is introduced into Schlemm's canal to scaffold open the canal
  Arms: OMNI canaloplasty and Hydrus with cataract surgery

SUMMARY:
The goal of this clinical trial is to look at the difference in pressure lowering effects in patients having two different combinations of minimally invasive glaucoma surgery (MIGS) at the time of their cataract surgery. Eligible patients will have mild to moderate glaucoma and be candidates for cataract surgery. The trial will look at the eye pressure before and one year after cataract surgery in patients. One eye in each patient will have cataract surgery with canaloplasty using OMNI. The patients other eye will have cataract surgery with canaloplasty and a HYDRUS stent. The trial will look at the differences in eye pressure and if patients are able to need fewer eye pressure lowering drops after surgery.

Study participants will undergo preop testing of pressure, vision, slit lamp exam, ocular coherence tomography (OCT) of the nerve fiber layer (NFL) analysis, and visual field prior to cataract surgery with MIGS. One day, one week, one month, 6 month, and 1 year exams will be performed to check pressure, vision, slit lamp exam, and number of necessary eye pressure medications in each eye.

DETAILED DESCRIPTION:
The purpose of this research study is to:

· Determine the differing pressure lowering effects between OMNI canaloplasty alone versus when combined with HYDRUS microstent. Both surgical study devices are widely used by themselves in conjunction with cataract surgery. While many surgeons have begun combining the two procedures, this will be one of the first studies to randomize (assign by chance) one eye to OMNI canaloplasty alone and the other eye to OMNI canaloplasty with HYDRUS stent and report the results after one year.

About 80 subjects aged 18 years and older will participate in this study.

WHAT WILL HAPPEN DURING THE STUDY?

Your participation in this study will last approximately one year and will include approximately seven study visits to the study center and two visits to the surgery center.

Screening:

Before any study-related tests and procedures are performed, you will be asked to read and sign this consent document. The following screening tests and procedures will then be performed to determine if you qualify to take part in this study:

* Visual field
* OCT analysis of the nerve and cornea - your nerve and cornea will be measured using optical coherence tomography (OCT) equipment. This is painless, non-invasive (it does not involve puncturing or cutting) and is similar to having photographs taken of your eye. You will be required to sit still during the brief scanning procedure (a few seconds)
* Slit lamp exam with gonioscopy - a close inspection of the front of the eye using a machine that magnifies the eye and provides a beam of light to light the structures of the eye
* Eye pressure test - measurement of the pressure inside the eye. The pressure in your eyes will be measured using an instrument known as a tonometer
* Visual acuity test - a test involving reading letters off a chart to determine how well you can see

This study will use competitive enrollment. This means that when a target number of subjects begins the study, all further enrollment will be closed. Therefore, it is possible that you could be

in the screening phase, ready to begin the study, and be discontinued without your consent if the target number of subjects has already begun the study.

If you qualify to take part in this study and go on to receive the study treatment, then the following will happen:

Washout Period: You will be asked to stop taking your eye drops to treat your glaucoma. This is called a washout period, during which the effects of these medications leave your body.

Study Treatment: You will be randomly assigned by chance (like the flip of a coin) to receive either OMNI canaloplasty or OMNI canaloplasty with HYDRUS microstent. You will have a 50% (1 in 2) chance of receiving OMNI canaloplasty alone or OMNI canaloplasty with HYDRUS microstent. This is a not a blinded study, which means that you, the study doctor, study staff and the sponsor will know the study treatment you are given.

You will have the following study visits and undergo the following procedures:

· Preoperative and postoperative care will be the same as a standard cataract surgery consisting of one day, one week, one month, six month and one year follow-up exams. The only difference for study subjects is they will be asked to stop all glaucoma drops one month prior to their pre-op exam and one year post-op exam.

After Study Treatment:

Glaucoma is a permanent and irreversible condition that requires lifelong monitoring with an eye care professional. Sometimes additional treatment is required. Your eye specialist will recommend follow-up care based on your personal findings.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with bilateral mild to moderate open angle glaucoma:

Including pseudoexfoliation (PXE) and pigment dispersion (PDS) According to ICD-10 guidelines and with visual field (VF) mean deviation -12 decibels (dB) or better With visually significant age-related cataract undergoing uncomplicated cataract surgery Able to randomize first eye to either treatment group, contralateral eye to receive other treatment Fairly symmetric glaucoma with cup to disc (C/D) asymmetry ≤ 0.1 and similar OCT RNFL and VF mean deviation IOP ≥ 20 mmHg and ≤ 36 mmHg after washout of ocular hypotensive medication(s); ≤3mmHg between the eyes Central corneal thickness (CCT) 480 to 620µm No prior ocular surgery including corneal refractive surgery; No selective laser trabeculoplasty (SLT) within 3 months of baseline visit, no history of intracameral implants Potential of good best corrected visual acuity at distance in the investigator's judgement of at least 0.1 LogMAR (20/25) postoperatively

Exclusion Criteria:

* Subjects with secondary glaucoma (traumatic, neovascular, mixed-mechanism, uveitic glaucoma) Uncontrolled intraocular pressure on maximum tolerated medical therapy; unable to wash-out intraocular pressure (IOP) lowering drops Anatomic exclusion of narrow anterior chamber angle (Shaffer grade I-II), other angle abnormalities leading to poor angle visualization H/o corneal disease or dystrophy Pathological myopia with degeneration that affects diagnostic imaging Clinically significant ocular pathology or degenerative diseases that affect vision, humphrey visual field (HVF), or OCT Inability to perform reliable HVF /OCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
change in unmedicated intraocular pressure from baseline at 12 months | 12 months
  check intraocular pressure at start date and at 12 months after washout of all pressure controlling drops

SECONDARY OUTCOMES:
reduction in number of medications needed to control intraocular pressure from baseline | 12 months
  compare number of drops prior to intervention with number of drops needed to control intraocular pressure at 12 months
percentage of patients with greater than 20% reduction in intraocular pressure from baseline | 12 months
  examine percentage of patients with a 20% reduction from their baseline unmedicated intraocular pressure at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McGraw, DO, Principal Investigator — Ridge Eye Care
Locations (4):
- United States (4):
  - Royo Eye Care, Marysville, California
  - Table Mountain Eye Care, Oroville, California
  - Ridge Eye Institute, Paradise, California
  - Feather River Eye Care, Yuba City, California

IPD SHARING:
Plan to Share IPD: No